CLINICAL TRIAL: NCT06420089
Title: CD5-deleted Chimeric Antigen Receptor Cells (Senza5 CART5) to Enhance Immunotherapy Against T Cell Non-Hodgkin Lymphoma (NHL): a First-in-human Phase I Clinical Trial
Brief Title: CD5-deleted Chimeric Antigen Receptor Cells (Senza5 CART5) for T Cell Non-Hodgkin Lymphoma (NHL)
Acronym: VIPER101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vittoria Biotherapeutics (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIPER 101
Record Dates: First submitted 2024-04-30; First posted 2024-05-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-07

CONDITIONS: T Cell Non-Hodgkin Lymphoma
Keywords: T Cell Lymphoma; Lymphoma; CD5KO CART5; Senza5 CART
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Senza5 CART5 with standard of care lymphodepletion (Experimental): Four treatment arms with Standard of Care Lymphodepletion:
  Fludarabine 25mg/m2 IV for 3 days Cyclophosphamide 250mg/m2 IV for 3 days
  Interventions: Drug: Senza5 CART5
- Senza5 CART5 without standard of care lymphodepletion (Experimental): Four treatment arms in patients are lymphopenic into the corresponding dose level.
  Interventions: Drug: Senza5 CART5

INTERVENTIONS:
Drug: Senza5 CART5 — The Senza5 CART5 drug product consists of a dual population of engineered autologous T cells: CD5 knockout (KO)cells and CD5KO-CART5 cells

SUMMARY:
This is an open-label phase I study to determine the safety and recommended phase 2 dose (RP2D) of Senza5 CART5 cells in patients with relapsed or refractory CD5 positive nodal T cell NHL. RP2D will be based on the safety, tolerability, pharmacokinetics, and preliminary efficacy of Senza5 CART5 cells. This trial will evaluate up to 5 dose levels using the Bayesian Optimal Interval (BOIN) design enrolling 3 patients in each cohort to assess safety and achieve therapeutic levels so that the RP2D of Senza5 CART5 cells given as a single IV infusion can be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed relapsed or refractory (r/r) CD5-positive nodal peripheral T-cell lymphoma (such as peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), nodal T-cell lymphomas with T-follicular helper (TFH) phenotype, including follicular T cell lymphoma, angioimmunoblastic lymphoma, or anaplastic large cell lymphoma) or other non-leukemic CD5+ aggressive mature T cell lymphomas (such as enteropathy-associated T cell lymphoma, monomorphic epitheliotropic intestinal T cell lymphoma, transformed mycosis fungoides, primary cutaneous aggressive epidermotropic CD8+ cytotoxic T-cell lymphoma, primary cutaneous insert gamma delta symbols lymphoma, or subcutaneous panniculitis like T cell lymphoma).
2. ≥50% expression of CD5 on flow cytometry or IHC on malignant cells on the most recent biopsy
3. Must have received at least one line of prior systemic therapy for their lymphoma; participants with anaplastic large cell lymphoma (ALCL) must have received prior brentuximab unless there was a contraindication to brentuximab.
4. Evaluable disease defined by at least one lesion that can be measured in least 1 dimension and measures at least 1.5 cm in its longest dimension by CT or PET scan, or bone/bone marrow involvement, or skin involvement.
5. No circulating CD5+ malignant cells identified by peripheral blood flow cytometry must be present.

Exclusion Criteria:

1. Pregnant or lactating (nursing) women.
2. HIV infection.
3. Concurrent use of systemic steroids or immunosuppressant medications.
4. Any uncontrolled active medical disorder that would preclude participation as outlined.
5. History of immunodeficiency.
6. History of prior chimeric antigen receptor therapy (CAR T), autologous or syngeneic HCT <100 days from transplant at the time of cell infusion or previous allo-HCT.
7. Active and/or systemic inflammatory or autoimmune diseases.
8. Signs or symptoms indicative of active CNS involvement.
9. Known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to lymphoma or previous lymphoma treatment.
10. Clinically apparent arrhythmia, or arrhythmias that are not stable on medical management
11. Current participation in or prior participation in a study of an investigational agent or using an investigational device within 2 weeks of the first dose of treatment.
12. Prior monoclonal antibody therapy within 4 weeks prior to study Day 1
13. Prior use of alemtuzumab
14. Prior chemotherapy targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1
15. Uncontrolled active infection requiring systemic therapy.
16. Circulating CD5+ malignant cells identified by peripheral blood flow cytometry present.
17. Active and/or systemic inflammatory or autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Determine the recommended phase 2 dose (RP2D) of Senza5 CART5 cells | 12 months
  Measure the occurrence of Dose Limiting Toxicity events of each dose level per arm

SECONDARY OUTCOMES:
Determine the safety of Senza5 CART5 cells | 12 months
  Quantify quantifying the type and frequency of adverse events
Determine the maximum tolerated dose (MTD) | 12 months
  Quantify the safety and tolerability of the highest dose
Determine the manufacturing feasibility of Senza5 CART5 | 12 months
  Quantify the number of product release failures and occurrence of dose failures (inability to meet targeted dose)
Determine efficacy of Senza5 CART5 | 12 months
  Measure the objective response rate
Determine efficacy of Senza5 CART5 | 12 months
  Measure the complete response rate
Determine efficacy of Senza5 CART5 | 12 months
  Measure the best overall response
Determine efficacy of Senza5 CART5 | 12 months
  Measure the duration of response
Determine efficacy of Senza5 CART5 | 12 months
  Measure the overall survival
Determine efficacy of Senza5 CART5 | 12 months
  Measure the progression free survival

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - University of Pennsylvania - Abramson Caner Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No